CLINICAL TRIAL: NCT02696577
Title: The Effect of Omega 3 on Pregnancy Complicated by Asymmetrical Intrauterine Growth Restriction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OIUGR
Record Dates: First submitted 2016-02-28; First posted 2016-03-02 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Intrauterine Growth Restriction
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Aspirin; Docosahexaenoic Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose aspirin (Active Comparator): Received aspirin 81mg once daily for 6 weeks
  Interventions: Drug: Low dose aspirin
- Low dose aspirin plus omega 3 group (Active Comparator): Received aspirin 81mg and omega 3 once daily for 6 weeks.
  Interventions: Drug: Low dose aspirin; Drug: Omega 3

INTERVENTIONS:
Drug: Low dose aspirin
Drug: Omega 3
  Arms: Low dose aspirin plus omega 3 group

SUMMARY:
Intrauterine growth restriction is a common and complex obstetric problem. Intrauterine growth restriction is noted to affect approximately 10-15 % of pregnant women. Intrauterine growth restriction is diagnosed antenatal; however, some of these fetuses, especially if unscreened during pregnancy, may be detected only in the neonatal period. It is very important for obstetricians and perinatologists to identify growth restricted fetuses, because this fetal condition is associated with significant perinatal morbidity and mortality.

Omega 3 is composed of polyunsaturated fatty acids with a double bond at the third carbon atom from the end of the carbon chain. The fatty acids have two ends, the carboxylic acid end, which is considered the beginning of the chain, thus "alpha", and the methyl end, which is considered the "tail" of the chain, thus "omega." Omega3 improve fetal wellbeing by two mechanisms: Firstly, maternal and docosahexaenoic acid supplementation during pregnancy and lactation normalizes intrauterine growth restriction induced changes in adipose deposition and visceral PPARγ expression. Secondly, maternal docosahexaenoic acid supplementation increases serum adiponectin, as well as adipose expression of adiponectin and adiponectin receptors. Novel findings suggest that maternal docosahexaenoic acid supplementation normalize adipose dysfunction and promote adiponectin-induced improvements in metabolic function in intrauterine growth restriction

ELIGIBILITY:
Inclusion Criteria:

* Age: from 20 - 35 years old.
* Pregnant from 30 week to 32 week gestation.
* Singleton pregnancy with asymmetrical intrauterine growth restriction .
* Normal uterine and umbilical Doppler indices at time of recruitment.

Exclusion Criteria:

* Multiple gestations.
* Hypertensive women.
* Premature rupture of membranes.
* Abnormal Doppler indices in the form of Doppler blood flow indices > 2 standard deviation , absent diastolic flow and lastly; reversed flow.
* Congenital fetal malformation.
* Pregnancy complicated by antepartum hemorrhage.
* Marked decrease in Amniotic fluid volume.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Estimated fetal weight (gm) | 1 year

SECONDARY OUTCOMES:
The changes in Doppler blood flow indices in both uterine arteries | 1 year
The changes in Doppler blood flow indices in umbilical artery | 1 year
Fetal weight at the time of delivery (gm) , | 1 year
Number of babies admitted to neonatal intensive care unit. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Ali MK, Amin ME, Amin AF, Abd El Aal DEM. Evaluation of the effectiveness of low-dose aspirin and omega 3 in treatment of asymmetrically intrauterine growth restriction: A randomized clinical trial. Eur J Obstet Gynecol Reprod Biol. 2017 Mar;210:231-235. doi: 10.1016/j.ejogrb.2017.01.002. Epub 2017 Jan 3. PMID 28068596